CLINICAL TRIAL: NCT01288885
Title: A Double-blind, Placebo-controlled, Dose Escalating Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Food-effect of Single Oral Doses of ASP1941 in Healthy Male Subjects
Brief Title: First in Men Study of Single Oral Doses of ASP1941 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 1941-CL-0001; 2006-002719-28 (EudraCT Number)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2011-02-03 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: ASP1941; Diabetes Mellitus; First in Men
MeSH Terms: conditions — Diabetes Mellitus | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ASP1941 — Oral
Drug: Placebo — Oral

SUMMARY:
This study determined the safety, tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of ASP1941 after a single oral dose (Part A). In addition, it was investigated whether the intake of food had an effect on the PK of ASP1941 (Part B).

DETAILED DESCRIPTION:
This study consists of two parts. Part A is a double-blind, placebo controlled single dose escalation study to evaluate the safety and tolerability of single ascending doses of ASP1941. Part B is an open label, crossover design food-effect study to evaluate the effect of fed conditions on the PK of ASP1941.

ELIGIBILITY:
Inclusion Criteria:

* Body weight between 60-100 kg, body mass index (BMI) between 20-30 kg/m2, inclusive

Exclusion Criteria:

* Fasting Plasma Glucose (FPG) > 6.4 mmol/l
* HbA1c > 6.2%
* Pulse <40 or >90 beats per minute; Systolic Blood Pressure (SBP) <90 or >140 mmHg; Diastolic Blood Pressure (DBP) <40 or >95mmHg

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2006-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability assessed by the incidence of adverse events, vital signs, physical examinations, 12-lead ECG and lab-tests | Up to 2 weeks after each administration

SECONDARY OUTCOMES:
Pharmacokinetics calculated by ASP1941 plasma concentration change | Up to 72 hours
Pharmacodynamics assessed by ASP1941 glucose concentration changes in blood and urine | Up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Manchester, United Kingdom